CLINICAL TRIAL: NCT00372125
Title: Nordic Study on the Effects of Growth Hormone (Norditropin SimpleXx) Treatment in Adults With Prader-Willi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Charlotte Hoeybye, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CH1234
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome; Growth hormone; Body composition
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norditropin SimpleXx (Active Comparator): 0.3 mg/day or 0.4 mg/day if bodyweight was below or above 100 kg,for 4 weeks, 0.6 mg/day or 0.8 mg/day, for 11 months.
  Interventions: Drug: Norditropin SimpleXx
- Placebo (Placebo Comparator): Placebo for 12 months
  Interventions: Drug: Norditropin SimpleXx

INTERVENTIONS:
Drug: Norditropin SimpleXx — 0.3-0.4 mg/day placebo or GH for 4 weeks. Thereafter 0.6-0.8 mg/day placebo or GH for 11 months. During the following 24 months open phase doses will be individually titrated.

SUMMARY:
The aim of this study is to study the effects of GH on body composition, lipid and glucose metabolism, physical performance and safety aspects in adults with PWS.The patients are randomized to either GH or placebo the first year of the study, subsequently followed by two years of GH treatment. the study is performed in Norway, Sweden and Denmark.

DETAILED DESCRIPTION:
OBJECTIVE(S):

Prader Willi syndrome (PWS) is a multi-symptomatic genetic disorder associated with abnormalities in the growth hormone (GH)-insulin-like-growth factor (IGF)-I axis and in the body composition. GH treatment is a registered indication in children with PWS, and improves growth rate and body composition. One pilot study in adult patients with clinical PWS has shown beneficial effects on body composition without simultaneous significant side effects. The aim of the present study is to evaluate the effects of GH treatment on body composition, muscle function and quality of life in PWS adults.

TRIAL DESIGN:

The study will be an investigator initiated and investigator sponsored multinational and multi-centre trial, including centres in Norway, Sweden and Denmark. Within each centre patients will be randomised (double blind) to one year treatment with daily injections of GH or placebo (efficacy), followed by a two year observation period on GH treatment (safety).

TRIAL POPULATION:

Twenty patients from each centre are included in the study. The patients need a genetically verified diagnosis and should be between 18 and 40 years old. Patients are excluded if GH treatment has been given within the last two years, if they have a malignancy or other serious diseases, in particular severe respiratory diseases.

ASSESSMENTS:

Effect is evaluated primarily as changes in body composition, activity of daily living and quality of life.

SAFETY: Before starting in the study all patients will be examined for tonsillary hypertrophy and sleep apnoea. Oral Glucose Tolerance Tests will be performed regularly.

TRIAL PRODUCT(S):

During the initial 4 weeks of the placebo-controlled study phase patients will be treated with sc injections of GH (Norditropin Simplexx) in the evening with doses of 0.3 mg/day respectively 0.4 mg/day if BW is below or above 100 kg. Thereafter doses will be increased to 0.6 mg/day (0.8 mg/day) and maintained fixed for 11 months. During the following 24 months open phase doses will be individually titrated.

ELIGIBILITY:
Inclusion Criteria:

* Genetically verified PWS diagnosis (by methylation and FISH test.)
* Between 18 and 50 years old
* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the treatment of the subject.)

Exclusion Criteria:

* Known or suspected allergy to GH preparation.
* Previous participation in this trial.
* GH treatment within the last 1 years
* Malignancy or other serious diseases (ex severe cardiovascular diseases, severe infections)
* Sexhormone treatment initiated within the last year
* Pregnancy
* Untreated respiratory impairment, untreated sleep apnoea or untreated respiratory infection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2005-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Changes in body composition (lean body mass and fat mass) measured by dual energy X-ray absorptiometry (DXA) | 36 months

SECONDARY OUTCOMES:
Bone mineral density measured by DXA | 36 months
Effects on forced expiratory volume (Peakflow) | 36 months
Standard photography appearance according to visual analogue scale (VAS) | 36 months
Effects on free and total IGF-I, IGF-binding protein (BP)-1 and 3 | 36 months
Effects on lipids (fasting triglycerides(TG), total, HDL and LDL cholesterol) | 36 months
Effects on body composition measured with bioimpedance | 36 months
Effects on haemoglobin (Hb), leucocyte and thrombocyte counts, FSH, LH, estradiol, Testosterone, inhibin B, TSH and Thyroxine | 36 months
Muscle and fat mass measured by abdominal and mid-femoral computerized tomography | 36 months
Activity of daily living measured a.m. Guralnik | 36 months
Quality of life estimated by questionnaires | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Hoybye, Dr., Principal Investigator — Department of Endocrinology and Diabetology, Karolinska Hospital; Jens S Christiansen, Professor, Study Chair — Århus University Hospital, Denmark
Locations (3):
- Center for rare Diseases, Department of Pediatrics, Skejby University Hospital, Aarhus N, Denmark
- Endokrinologisk seksjon, Med Avd, Rikshospitalet, Oslo, Norway
- Department of Endocrinology and Diabetology, Karolinska Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Shukur HH, Hussain-Alkhateeb L, Farholt S, Norregaard O, Jorgensen AP, Hoybye C. Effects of Growth Hormone Treatment on Sleep-Related Parameters in Adults With Prader-Willi Syndrome. J Clin Endocrinol Metab. 2021 Aug 18;106(9):e3634-e3643. doi: 10.1210/clinem/dgab300. PMID 33950234
- [Derived] Olarescu NC, Jorgensen AP, Godang K, Jurik AG, Froslie KF, Bollerslev J. Dual-energy X-ray absorptiometry is a valid method to estimate visceral adipose tissue in adult patients with Prader-Willi syndrome during treatment with growth hormone. J Clin Endocrinol Metab. 2014 Sep;99(9):E1727-31. doi: 10.1210/jc.2014-2059. Epub 2014 Jun 23. PMID 24955611
- [Derived] Jorgensen AP, Ueland T, Sode-Carlsen R, Schreiner T, Rabben KF, Farholt S, Hoybye C, Christiansen JS, Bollerslev J. Glucose homeostasis in adults with Prader-Willi syndrome during treatment with growth hormone: results from a 12-month prospective study. Growth Horm IGF Res. 2014 Feb;24(1):16-21. doi: 10.1016/j.ghir.2013.11.002. Epub 2013 Dec 4. PMID 24360789
- [Derived] Jorgensen AP, Ueland T, Sode-Carlsen R, Schreiner T, Rabben KF, Farholt S, Hoybye C, Christiansen JS, Bollerslev J. Two years of growth hormone treatment in adults with Prader-Willi syndrome do not improve the low BMD. J Clin Endocrinol Metab. 2013 Apr;98(4):E753-60. doi: 10.1210/jc.2012-3378. Epub 2013 Feb 22. PMID 23436915